CLINICAL TRIAL: NCT06916702
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Rising Oral Doses of BI 3031185 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Different Doses of BI 3031185 Are Tolerated by Healthy Men
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1516-0002; 2024-516921-29-00 (Registry Identifier: CTIS (EU)); U1111-1311-3555 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-03-27; First posted 2025-04-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors may be unblinded upon request, except for Electrocardiogram (ECG) laboratory staff, who shall remain blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose group 1 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo
- Dose group 2 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo
- Dose group 3 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo
- Dose group 4 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo
- Dose group 5 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo
- Dose group 6 (receiving BI 3031185 or Placebo, plus midazolam) (Experimental)
  Interventions: Drug: BI 3031185; Drug: Midazolam; Drug: Placebo

INTERVENTIONS:
Drug: BI 3031185 — BI 3031185
Drug: Midazolam — Midazolam
Drug: Placebo — Placebo matching BI 3031185

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 3031185 in healthy male subjects following administration of multiple rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body Mass Index (BMI) of 20.0 to 29.9 kg/m (inclusive) and body weight of at least 60 kg
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, Pulse rate (PR) or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement at screening of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 50 to 89 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | Up to Day 54

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 3031185 in plasma at steady state over a uniform dosing interval τ ((AUC) τ,ss ) | Up to Day 42
Maximum measured concentration of BI 3031185 in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | Up to Day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com